**Protocol Number:** 20160370

**Date:** 12 June 2020 

## Statistical Analysis Plan

| Protocol Title: | A Phase 1b Multicenter, Op<br>Study to Assess the Safety<br>AMG 420 as Monotherapy i<br>Relapsed and/or Refractory | and Efficacy of<br>n Subjects With<br>Multiple Myeloma |
|---|---|---|
| Short Protocol Title: | A Phase 1b Study to Assess AMG 420 Monotherapy in Subjects with Relapsed and/or Refractory Multiple Myeloma | |
| Protocol Number: | 20160370 | |
| NCT Number: | NCT03836053 | |
| Authors: | | |
| | Biostatistician II, IQVIA | |
| | Biostatistics Director, Amgen Inc | |
| Sponsor: | Amgen Inc | |
| | One Amgen Center Drive<br>Thousand Oaks, CA 91320 | |
| SAP Date: | <b>Document Version</b> | <u>Date</u> |
| | Amendment 1 (v[2.0]) | 12 June 2020 |



**Protocol Number:** 20160370

**Date:** 12 June 2020 

| Version Number | Date<br>(DDMMMYYYY) | Summary of Changes, including rationale for changes |
|---|---|---|
| Original (v1.0) | 11JAN2019 | NA |
| Amendment 1 (v2.0) | 12Jun2020 | Removal of Phase 1b Part 2 (combination cohort) and Phase 2 text globally |



**Protocol Number:** 20160370

**Date:** 12 June 2020

#### **Table of Contents**

| rabio | e of Co | ntents | 3 |
|---|---|---|---|
| 1. | Introdu | uction | 9 |
| 2. | Object | tives, Endpoints and Hypotheses | 9 |
| | 2.1 | Objectives and Endpoints | |
| | 2.2 | Hypotheses and/or Estimations | |
| 3. | Study | Overview | 11 |
| | 3.1 | Study Design | 11 |
| | 3.2 | Sample Size | 13 |
| | 3.3 | Adaptive Design | 13 |
| 4. | Covari | iates and Subgroups | 13 |
| | 4.1 | Planned Covariates | 13 |
| | 4.2 | Subgroups | 13 |
| 5. | Definit | ions | 14 |
| 6. | Analys | sis Sets | 20 |
| | 6.1 | Safety Analysis Set | 20 |
| | 6.2 | Dose Limiting Toxicity Evaluable Analysis Set | 20 |
| | 6.3 | Pharmacokinetic/Pharmacodynamic Analyses Set(s) | 20 |
| | 6.4 | Retreatment Analysis Set | 21 |
| 7. | Planne | ed Analyses | 21 |
| | 7.1 | Interim Analysis and Early Stopping Guidelines | 21 |
| | | 7 4 4 Interior Analysis | |
| | | 7.1.1 Interim Analyses | 21 |
| | | 7.1.1 Interim Analyses | |
| | 7.2 | · | 21 |
| | 7.2<br>7.3 | 7.1.2 Dose Level Review Team | 21<br>21 |
| 8. | 7.3 | 7.1.2 Dose Level Review Team | 21<br>21<br>21 |
| 8. | 7.3 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis | 21<br>21<br>21 |
| 8. | 7.3<br>Data 9 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance | 21<br>21<br>21<br>21 |
| 8. | 7.3<br>Data 9<br>8.1 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance General Principles | 21<br>21<br>21<br>21<br>21 |
| 8. | 7.3<br>Data 8<br>8.1<br>8.2 | 7.1.2 Dose Level Review Team. Primary Analysis Final Analysis Screening and Acceptance. General Principles Data Handling and Electronic Transfer of Data | 21<br>21<br>21<br>21<br>21<br>21 |
| 8. | 7.3<br>Data 5<br>8.1<br>8.2<br>8.3 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance General Principles Data Handling and Electronic Transfer of Data Handling of Missing and Incomplete Data | 21<br>21<br>21<br>21<br>21<br>21 |
| 8. | 7.3<br>Data 8<br>8.1<br>8.2<br>8.3<br>8.4 | 7.1.2 Dose Level Review Team. Primary Analysis Final Analysis Screening and Acceptance. General Principles Data Handling and Electronic Transfer of Data Handling of Missing and Incomplete Data Detection of Bias | 21<br>21<br>21<br>21<br>21<br>21<br>22 |
| 8. | 7.3<br>Data 5<br>8.1<br>8.2<br>8.3<br>8.4<br>8.5 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance General Principles Data Handling and Electronic Transfer of Data Handling of Missing and Incomplete Data Detection of Bias Outliers | 21<br>21<br>21<br>21<br>21<br>21<br>22<br>22 |
| <ol> <li>8.</li> <li>9.</li> </ol> | 7.3 Data S 8.1 8.2 8.3 8.4 8.5 8.6 8.7 Statist | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance General Principles Data Handling and Electronic Transfer of Data Handling of Missing and Incomplete Data Detection of Bias Outliers Distributional Characteristics Validation of Statistical Analyses ical Methods of Analysis | 21<br>21<br>21<br>21<br>21<br>21<br>22<br>22 |
| | 7.3 Data S 8.1 8.2 8.3 8.4 8.5 8.6 8.7 Statist 9.1 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance. General Principles Data Handling and Electronic Transfer of Data Handling of Missing and Incomplete Data Detection of Bias Outliers Distributional Characteristics Validation of Statistical Analyses ical Methods of Analysis General Considerations | 21<br>21<br>21<br>21<br>21<br>22<br>22<br>22<br>22 |
| | 7.3 Data S 8.1 8.2 8.3 8.4 8.5 8.6 8.7 Statist 9.1 9.2 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance General Principles Data Handling and Electronic Transfer of Data Handling of Missing and Incomplete Data Detection of Bias Outliers Distributional Characteristics Validation of Statistical Analyses ical Methods of Analysis. General Considerations Subject Accountability | 21<br>21<br>21<br>21<br>21<br>22<br>22<br>22 |
| | 7.3 Data S 8.1 8.2 8.3 8.4 8.5 8.6 8.7 Statist 9.1 | 7.1.2 Dose Level Review Team Primary Analysis Final Analysis Screening and Acceptance. General Principles Data Handling and Electronic Transfer of Data Handling of Missing and Incomplete Data Detection of Bias Outliers Distributional Characteristics Validation of Statistical Analyses ical Methods of Analysis General Considerations | 21<br>21<br>21<br>21<br>21<br>22<br>22<br>22<br>22<br>22<br>22 |



**Protocol Number:** 20160370

| Date: | 12 June 2020 |
|-------|--------------|

| | 9.5 | Efficacy | / Analyses | | 24 |
|---|---|---|---|---|---|
| | | 9.5.1 | Analyses | of Key Secondary Efficacy Endpoint(s) | 24 |
| | | | 9.5.1.1 | Overall Response Rate | 24 |
| | | | 9.5.1.2 | Duration of Response | 24 |
| | | | 9.5.1.3 | MRD Negativity at CR | 24 |
| | | 9.5.2 | Analyses | of Secondary Efficacy Endpoint(s) | 24 |
| | | | 9.5.2.1 | Progression-free Survival | 24 |
| | | | 9.5.2.2 | Overall Survival | 24 |
| | | | 9.5.2.3 | Time to Response | |
| | | 9.5.3 | Analyses | of Exploratory Efficacy Endpoint(s) | 2 |
| | 9.6 | Safety A | Analyses | | 2 |
| | | 9.6.1 | Analyses | of Safety Endpoint(s) | 2 |
| | | 9.6.2 | Adverse | Events | 2 |
| | | 9.6.3 | Laborato | ry Test Results | 27 |
| | | 9.6.4 | Vital Sigr | ns | 27 |
| | | 9.6.5 | Physical | Measurements | 28 |
| | | 9.6.6 | Electroca | ırdiogram | 28 |
| | | | | | 28 |
| | | 9.6.8 | | e to Investigational Product | |
| | | 9.6.9 | Exposure | e to Concomitant Medication | 28 |
| | 9.7 | Other A | Analyses | | 29 |
| | | 9.7.1 | • | ses | 29 |
| | | 9.7.2 | | of Pharmacokinetic or okinetic/Pharmacodynamic Endpoints | 29 |
| | | 9.7.3 | Analyses | of Clinical Outcome Assessments | 29 |
| | | 9.7.4 | Analyses | of Health Economic Endpoints | 29 |
| | | 9.7.5 | Analyses | of Biomarker Endpoints | 29 |
| 10. | Chan | ges From | Protocol-sp | pecified Analyses | 29 |
| 11. | Litera | ture Citat | ions / Refer | ences | 30 |
| 12. | Priori | tization of | Analyses | | 3 |
| 13. | Data | Not Cove | red by This | Plan | 3′ |
| 14. | Appe | ndices | | | 32 |
| | Appe | ndix A. R | Reference Va | alues/Toxicity Grades | 33 |
| | Appe | ndix B. G | Guidance for | Response Confirmation | 3 |
| | Appe | ndix C. C | Clinical Outco | ome Assessment Forms/Instruments | 37 |
| | Appe | ndix D. H | lealth Econo | omic Forms/Instruments | 38 |
| | Appe | ndix E. D | etails of PK | or PK/PD Methods for Modeling | 39 |



**Protocol Number:** 20160370

**Date:** 12 June 2020 

#### **List of Tables**

| Table 1. | Rules for Holding Enrollment in Phase 1b | 12 |
|----------|-------------------------------------------|----|
| Table 2. | Conventions for Censoring for PFS and DOR | 17 |



**Protocol Number:** 20160370

**Date:** 12 June 2020 

## **List of Abbreviations and Definition of Terms**

| Abbreviation or Term | Definition/Explanation |
|---|---|
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| APRIL | a proliferation-inducing ligand |
| AST | aspartate aminotransferase |
| AUC <sub>last</sub> | area under the concentration-time curve from time 0 to the last measurable concentration |
| BAFF | B-cell activating factor |
| BAFF-R | B-cell activating factor receptor |
| BiTE® | bispecific T-cell engager |
| ВМ | bone marrow |
| BOR | best overall response |
| CAR | chimeric antigen receptor |
| cIV | continuous intravenous |
| C <sub>max</sub> | maximum concentration |
| CR | complete response |
| Css | steady-state concentration |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DLRM | dose level review meeting |
| DLRT | dose level review team |
| DLT | dose limiting toxicity |
| DOR | duration of response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EM | Extramedullary |
| EOI | end of infusion |
| EOS | end of study |
| EOT | end of treatment |
| FDA | Food and Drug Administration |
| FIH | first-in-human |
| FISH | fluorescent in situ hybridization |



**Protocol Number:** 20160370

**Date:** 12 June 2020 

| A | |
|---|---|
| Abbreviation or Term | Definition/Explanation |
| FLC | free light chain |
| IMiD | Immunomodulator |
| IMWG | International Myeloma Working Group |
| ISS | International Staging System |
| IV | intravenous(ly) |
| KM | Kaplan-Meier |
| LTFU | long-term follow-up |
| MR | minimal response |
| MRD | minimal residual disease |
| MTD | maximum tolerated dose |
| mTPI | modified toxicity probability interval |
| ORR | overall response rate |
| os | overall survival |
| PD | progressive disease |
| PFS | progression-free survival |
| PI | proteasome inhibitor |
| PK | pharmacokinetic(s) |
| PR | partial response |
| PR interval | PR interval is measured from the beginning of the P wave to the beginning of the QRS complex in the heart's electrical cycle as measured by ECG or partial response |
| QRS interval | QRS interval is the interval between the Q wave and the S wave in the heart's electrical cycle as measured by ECG; represents the time it takes for the depolarization of the ventricles |
| QTc interval | QT interval corrected for heart rate using accepted methodology |
| RRMM | Relapsed and/or refractory multiple myeloma |
| SC | subcutaneous(ly) |
| sCR | stringent complete response |
| sFLC | serum free light chain |
| SFU | safety follow-up |
| SPEP | serum protein electrophoresis |
| t <sub>1/2</sub> | half-life |
| TBL | total bilirubin |
| TFI | treatment-free interval |
| TLS | tumor lysis syndrome |



**Protocol Number: 20160370** 

**Date:** 12 June 2020 

| Abbreviation or Term | Definition/Explanation |
|------------------------|-------------------------------|
| TNF | tumor necrosis factor |
| TPI | toxicity probability interval |
| T <sub>reg</sub> cells | regulatory T cells |
| UIFE | urine immunofixation |
| ULN | upper limit of normal |
| UPEP | urine protein electrophoresis |
| US | United States |
| VGPR | very good partial response |



Protocol Number: 20160370

**Date:** 12 June 2020 

#### 1. Introduction

The purpose of this Statistical Analysis Plan (SAP) is to provide details of the statistical analyses that have been outlined within the protocol **amendment 4** for study 20160370, AMG 420 dated **20 May 2020**. The scope of this plan includes the interim analysis, primary analysis and final analysis that are planned and will be executed by the Amgen Global Biostatistical Science department unless otherwise specified.

## 2. Objectives, Endpoints and Hypotheses

## 2.1 Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Phase 1b | |
| Primary | |
| <ul> <li>Establish the safety and<br/>tolerability of AMG 420 at dose<br/>levels of 400 μg/day and 600<br/>μg/day in subjects with relapsed<br/>and/or refractory multiple<br/>myeloma (RRMM)</li> </ul> | Dose-limiting toxicities (DLTs),<br>treatment-emergent adverse<br>events, treatment-related adverse<br>events and changes in vital signs,<br>electrocardiograms (ECGs), and<br>clinical laboratory tests |
| Key Secondary | |
| Estimate overall response rate (ORR) and duration of response (DOR) of AMG 420 in subjects with RRMM | ORR DOR |
| Evaluate the rate of minimal residual<br>disease (MRD)-negativity at the time<br>of CR | MRD negativity at the time of CR |
| Secondary | |
| Establish the safety and tolerability of<br>AMG 420 in subjects with<br>extramedullary relapsed multiple<br>myeloma | DLTs, treatment-emergent adverse<br>events, treatment-related adverse<br>events, and changes in vital signs,<br>ECGs, and clinical laboratory tests |
| Characterize the pharmacokinetics<br>(PK) of AMG 420 when administered<br>as 4-week continuous intravenous<br>(cIV) infusion | AMG 420 PK parameters including,<br>but not limited to, half-life (t <sub>1/2</sub> ),<br>clearance, and apparent C <sub>ss</sub> |
| Evaluate other measures of<br>anti-myeloma activity of AMG 420 in<br>subjects with RRMM: | Efficacy parameters according to<br>International Myeloma Working Group<br>(IMWG) response criteria, per<br>investigator assessment: |



Protocol Number: 20160370 Date: 12 June 2020 

| Objectives | Endpoints |
|---|---|
| Secondary (Continued) | |
| <ul> <li>Time to response</li> <li>Progression-free survival (PFS)</li> <li>Overall survival (OS)</li> <li>Best overall response (BOR)</li> </ul> | <ul><li>Time to response</li><li>PFS</li><li>OS</li><li>BOR</li></ul> |
| Exploratory for Phase1b | |
| Enter Exploratory Objectives Endpoints | |

Protocol Number: 20160370

**Date:** 12 June 2020 

#### 2.2 Hypotheses and/or Estimations

The ORR according to IMWG response criteria along with 95% CI will be calculated per **investigator** assessment for subjects with RRMM. The lower bound of the binomial 2-sided 95% confidence interval for ORR not lower than 35% is considered clinically meaningful.

#### 3. Study Overview

#### 3.1 Study Design

This is a phase 1b, multicenter, non-randomized, open-label expansion study. AMG 420 will be evaluated in adult subjects with RRMM.

The study will consist of up to a 21-day screening, a treatment, safety follow-up (SFU), and long-term follow-up (LTFU) period. In the treatment period, treatment will be continued until progressive disease (PD) or relapse as defined by IMWG response criteria, unacceptable safety events, next anti-multiple myeloma treatment, or other reason for permanent treatment discontinuation. All subjects will be assessed for anti-myeloma activity according to the IMWG response criteria. An SFU visit will be conducted 30 (+3) days after last administration of AMG 420, and an LTFU period that will begin after the SFU visit is completed. The total duration of the LTFU will be up to 5 years from the first dose of AMG 420 as described in Study Schema of protocol section 2.1.

#### Phase 1b (Monotherapy Dose Confirmation)

In phase 1b, approximately 10 subjects will be treated at the 400  $\mu$ g/day dose (comprising cohort 1). Approximately 10 subjects will be treated at the 600  $\mu$ g/day dose level (cohort 2). Each subject in phase 1b will have at least a 30-day SFU.



Protocol Number: 20160370

**Date:** 12 June 2020 

The dose level review team (DLRT) will **convene and** review all available safety, laboratory, and pharmacokinetic (PK) data at the following scheduled time points:

 After at least 10 subjects in cohort 1 (400 μg/day dose level) in phase 1b have had the opportunity to complete the 4-week infusion period of the first treatment cycle: On the basis of this review, the DLRT will make a recommendation regarding the initiation of the 600 μg/day dose level (cohort 2) in phase 1b.

- After at least 3 subjects with extramedullary (EM) relapsed disease in cohort 1 (400 μg/day dose level) have had the opportunity to complete the 4-week infusion period of the first treatment cycle: On the basis of this review, the DLRT will make a recommendation regarding the appropriateness of continued enrollment of subjects with EM relapsed disease to cohort 2 in phase 1b (600 μg/day dose level). Please note that enrollment of subjects with EM relapsed disease to cohort 2 in phase 1b will not be allowed until this safety review of the first 3 subjects with EM disease is completed by the DLRT.
- After the first 3 subjects have been dosed with AMG 420 at 600  $\mu g$ /day for the full 4-week infusion cycle.

The safety data will be reviewed on an ongoing basis and enrollment may be terminated at any time. To further reduce the risk of overdose to ongoing and future subjects, protocol-defined enrollment holding rules will be used. These rules are based on a modified Toxicity Probability Interval (mTPI), where the target Toxicity Probability Interval (TPI) is a dose-limiting toxicity (DLT) probability from 20% to 33% and the overdose TPI is > 33% DLT probability. Enrollment to the ongoing dose level/schedule will be paused per the following rules during enrollment into phase 1b cohort 1 and 2.

Table 1. Rules for Holding Enrollment in Phase 1b

| Number of DLTs | ≥ 2 | ≥ 3 | ≥ 4 |
|----------------------------|-----|-----|-----|
| Number of Treated Subjects | ≤ 4 | ≤ 6 | ≤ 8 |

If the rules for pausing enrollment are met, no further enrollment to the respective dose level/schedule will be allowed until after a careful review of all safety data by the DLRT. Additionally, enrollment will not resume until the protocol has been amended to include additional safeguards for subject safety (eg, modifications to dose level and schedule).

Subjects with EM disease will be able to enroll into cohort 2 **after** the safety evaluation is complete for 3 subjects with EM disease treated at 400 µg/day (cohort 1).

An **investigator** will review efficacy data and assess outcomes in accordance with IMWG criteria. **Investigator** assessments will be used for efficacy analysis.



Protocol Number: 20160370

**Date:** 12 June 2020 

## 3.2 Sample Size

Approximately 20 subjects will be enrolled in this study.

#### 3.3 Adaptive Design

The rules for halting enrollment are based on an mTPI design. The mTPI models the probability of toxicity for each dose level using a Bayesian model where each dose level has the same prior on the probability of toxicity, a Beta (1,1). When subjects are treated at the current dose level, the posterior probability of toxicity is updated using the observed data from this level. Enrollment recommendations are made based on this posterior probability of toxicity, using three toxicity probability intervals (TPI).

- Under-dosing TPI: DLT rate from 0 to < 20%</li>
- Target TPI: DLT rate from 20% to 33%
- Over-dosing TPI: DLT rate > 33%

For the current dose level and after adjusting for the width of each TPI interval, if the DLT rate is most likely in the under-dosing TPI or most likely in the target TPI then the recommendation is to continue enrollment at the current level. If the DLT rate is most likely in the over-dosing TPI then the recommendation is to halt enrollment.

#### 4. Covariates and Subgroups

#### 4.1 Planned Covariates

There are no planned covariates in this study.

#### 4.2 Subgroups

The baseline variables for the subgroup analyses may include:

- baseline demographics and characteristics:
  - age (< 65, 65-74, ≥ 75 years)</li>
  - sex (female, male)
  - race (White, Asian, other)
- baseline disease characteristics:
  - revised International Staging System (ISS) stage (Stage I, Stages II or III)
  - BM percent of plasma cells (< 50%, ≥ 50%)</li>
  - \_ \_
  - extramedullary disease (yes, no). Until safety evaluation is complete for 3 subjects with EM disease, imaging evaluation at screening will be used to document EM disease status.
- number of prior lines of therapy (only 3, > 3)



Protocol Number: 20160370

**Date**: 12 June 2020 

- prior allogeneic HSCT (yes, no)
- refractory to
  - IMiD (yes, no)
  - PI (yes, no)
  - IMiD + PI (yes, no)
  - daratumumab or other CD 38-targeting antibody (yes, no)

Subgroup analysis will not be performed due to each sub group may not have justifiable count as less number of sample size.

#### 5. Definitions

#### Adverse Event (AE)

An adverse event is defined as any untoward medical occurrence in a clinical trial subject. The event does not necessarily have a causal relationship with study treatment. The definition of adverse events includes worsening of a preexisting medical condition. A preexisting condition that has not worsened during the study, or involves an intervention, is not considered an adverse event.

#### Age at Enrollment

Subject age at enrollment will be determined using the age in years reported in the clinical database.

#### <u>Baseline</u>

For any variable, unless otherwise specified the baseline is the last assessment taken prior to the first administration of AMG 420. For parameters/assessments not scheduled to be performed (or scheduled but not performed) on the same day as the first administration of AMG 420, the baseline value is the value from the screening period measured closest to the day of first administration of AMG 420.

#### Baseline ECG Values in Triplicate

For the three sets of triplicate pre-dose ECG, the mean of values in a triplicate should be calculated before taking the mean of the three sets of averages. For all post-baseline ECG, the mean value for measurements taken at the same assessment will be calculated and used in the analysis. When an ECG is missing within a triplicate, all available data will be averaged for that time point.



Protocol Number: 20160370

**Date:** 12 June 2020 

#### Death Date

For subjects who die during the study, the death date will be recorded on the end of study CRF in the date subject ended study field. Incomplete death dates where only the day of death date is missing will be imputed using the following rules:

Day 1 of the month will be used if year and month indicate that death happened in different month from last known alive date;

One day after last known alive date will be used if death happened in the same month as last known alive date.

The imputed death date will be used in calculation of duration of response, progressionfree survival and overall survival.

#### **Dose-limiting Toxicities (DLTs)**

Investigators determine whether a TEAE qualifies as a DLT per the definition described in protocol Section 7.4.1. For an adverse event to qualify as a DLT, the start date must be within 28 days from the date of the first dose of investigational product.

#### Best Overall Response

Best overall response for a subject is the best observed post baseline disease response per the International Myeloma Working Group Uniform Response Criteria for Multiple Myeloma (IMWG-URC). **The detailed algorithm is provided in** Appendix B.

#### Overall Response Rate (ORR)

ORR refers to the proportion of subjects with an objective response. Objective response refers to any of the following responses per the International Myeloma Working Group Uniform Response Criteria for Multiple Myeloma (IMWG-URC): (sCR, CR, VGPR or PR) Per IMWG-URC, any response requires 2 consecutive assessments made any time before starting any new therapy. Subjects who do not experience a sCR/CR/VGPR/PR or do not have any follow-up tumor assessments will be regarded as non-responders.

#### Duration of Response (DOR)

Duration of response (DOR) will be calculated for subjects who achieve a PR or better. For such subjects, the duration of overall response is defined as the time (months) from first documentation of response to disease progression or death due to any cause. Dates of progression and censoring will be determined as described for the analysis of PFS.



Protocol Number: 20160370

**Date:** 12 June 2020 

DOR (in months) = (Earliest date of disease progression, death, censor - Date of first observation of PR or better before confirmation + 1)/30.4

Subjects who have not ended their response at the time of analysis will have DOR censored on the date of their latest evaluable assessment.

#### Time to response

Time to response applies for subjects who achieved best overall response of PR, VGPR, CR or sCR. Time to response is calculated as the number of months (one mont = 30.4 days) from the first administration of AMG 420 to the first objective assessment of response (ie, date of the first detection of response) as per IMWG-URC.

TTR (in months) = (Date of objective response – Date of first dose + 1)/30.4

#### MRD Negativity (MRD-)

MRD- is defined as a response of CR or sCR accompanied by any of the following types of MRD negativity.

- Sustained MRD-
- Sequencing MRD-
- Imaging plus MRD-

Subjects who do not experience a MRD negativity or do not have any evaluable followup assessments will be regarded as MRD non-responders.

#### Progression-free survival (PFS)

Progression free survival (PFS) is defined as number of months between start of treatment and first evidence of documented disease progression or death (due to any cause), whichever occurs first.

PFS (in months) = (Earliest date of disease progression, death, censor – Date of first dose + 1)/30.4

Progression-free survival will be right-censored for subjects who meet one of the following conditions: 1) no post baseline disease assessments, 2) non-protocol systemic anticancer treatment started before documentation of PD or death, 3) death or disease progression after more than 1 missed disease assessment visit or 4) alive and does not have documentation of PD before a data analysis cutoff date. For such subjects, the



Protocol Number: 20160370

**Date:** 12 June 2020 

primary analysis of PFS will be right-censored according to the conventions described in Table 2.

Table 2. Conventions for Censoring for PFS and DOR

| Situation | Date of Progression or Censoring | Outcome |
|---|---|---|
| No post baseline disease assessments** | Date of first dose | Censored |
| New anticancer therapy started before documentation of PD or death | Date of last evaluable disease assessment prior to start of new anticancer therapy | Censored |
| Death or PD immediately after more than 1 consecutively missed disease assessment visit* | Date of last evaluable disease assessment visit before the first missed visit | Censored |
| Alive and without PD documentation (including lost to follow-up without PD) | Date of last evaluable disease assessment | Censored |
| Death or PD between planned disease assessments | Date of death or first disease assessment showing PD, whichever occurs first | Progressed |
| Death before first disease assessment | Date of death | Progressed |

<sup>\*</sup> If death or PD is more than 84 days after previous disease assessment, or Study Day 1 if there is no previous disease assessment.

#### Overall survival (OS)

Overall survival is defined as the interval from Study Day 1 until death due to any cause; otherwise, OS is censored on the last recorded date on which the subject was alive.

#### Last Evaluable Disease Assessment Date

For responses assessed by investigator, last disease assessment date is the last evaluable response assessment date collected using IMWG Response CRF (except the response assessment date of Inevaluable) before confirmed PD, on or before new anticancer therapies or procedures.

#### Last Known Alive Date

For subjects not known to have died, their last date known to be alive will be determined as the latest date associated with clinic visits before data cutoff date including, for example, but not limited to the following:

- Date of Enrollment on Subject Enrollment CRF
- Date First Taken, Date Last Taken on Concomitant Medications CRF



<sup>\*\*</sup> Only apply to PFS.

Protocol Number: 20160370

**Date**: 12 June 2020 

 Date Performed on ECOG Performance Status, Vital Signs, Electrocardiogram, Procedures CRFs

- Admission Date, Discharge Date on Hospitalizations CRF
- Date of Examination on Physical Measurement CRF
- Date Collected on Reproductive Status and Pregnancy Test (Local Lab), Chemistry (Local Lab), Hematology (Local Lab), Coagulation (Local Lab), Urinalysis (local Lab), Immunology (Local lab) CRFs and in central lab data
- Date of Assessment on IMWG Response for Time Point, Peripheral Neuropathy Assessment CRFs
- Start Date and End Date on Investigational Product Administration CRF
- Date Started and Date Ended or Resulted in Death on Events CRF
- Start date, Stop date on Anti-Myeloma / Anti-Cancer Therapies, Other Protocol Required Therapy (GLUCOCORTICOID), Other Protocol Required Therapy (Tocilizumad), Hematopoietic Stem Cell Transplantation Autologous, Hematopoietic Stem Cell Transplantation Allogenic CRFs
- Subject Status Date if status is Alive on Survival Status CRF
- Assessment Date on Skeletal Survey and Plasmacytoma Assessment CRF
- End\_of study date if the subject's primary reason for ending study is not "Lost to follow-up"

#### Fridericia-corrected QT Interval (QTcF)

The Fridericia correction will be calculated from the investigator reported QT (msec) and RR interval (msec), as follows:

 $QTcF=QT/(RR/1000)^{1/3}$ 

#### Change From Baseline

Change from Baseline is the arithmetic difference between post-dose assessments and Baseline value.

Change (absolute) from Baseline = (Post-baseline Value – Baseline Value)

Change (percent) from Baseline

= [(Post-baseline Value – Baseline Value)/Baseline Value] x 100

#### Investigational Product (IP)

The term 'investigational product' is used in reference to AMG 420.

#### Primary Completion:

The primary completion date is defined as the date when the last subject is assessed or receives an intervention for the final collection of data for the primary endpoint(s), for the



Protocol Number: 20160370

**Date:** 12 June 2020 

purposes of conducting the primary analysis, whether the study concluded as planned in the protocol or was terminated early.

If the study concludes prior to the primary completion date originally planned in the protocol (ie, early termination of the study), then the primary completion will be the date when the last subject is assessed or receives an intervention for evaluation in the study (ie, last subject last visit).

#### End of Study

The end of study (EOS) date is defined as the date when the last subject across all sites is assessed or receives an intervention for evaluation in the study (ie, last subject last visit), following any additional parts in the study (eg, LTFU), as applicable.

#### Lost to Follow-up

A subject will be considered lost to follow-up if he or she repeatedly fails to return for scheduled visits and is unable to be contacted by the study site. The following actions must be taken if a subject fails to return to the clinic for a required study visit:

- The site must attempt to contact the subject and reschedule the missed visit as soon as possible and counsel the subject on the importance of maintaining the assigned visit schedule and ascertain whether or not the subject wishes to and/or is able to continue in the study.
- In cases in which the subject is deemed lost to follow-up, the investigator or designee must make every effort to regain contact with the subject (where possible, 3 telephone calls and, if necessary, a certified letter to the subject's last known mailing address or local equivalent methods). These contact attempts are to be documented in the subject's medical record.
- If the subject continues to be unreachable, he/she will be considered to have withdrawn from the study with a primary reason of lost to follow-up.
- For subjects who are lost to follow-up, the investigator can search publicly available records where permitted to ascertain survival status. This ensures that the data set(s) produced as an outcome of the study is/are as comprehensive as possible.

#### Study Day

Post study day: study day= (date - date of Study Day 1) + 1

Pre study day: study day= (date – date of Study Day 1)

#### Study Day 1

It is defined as the first day that protocol-specified investigational product is administered to the subject.



Protocol Number: 20160370

**Date:** 12 June 2020 

#### <u>Treatment-emergent Adverse Event (TEAE)</u>

A treatment-emergent adverse event is any adverse event starting on or after the first administration of investigational product, as determined by the flag indicating if the adverse event started prior to the first dose on the Events CRF, and up to and including 33 days after the last IP dose date or EOS date, whichever occurs first. The severity of each adverse event will be graded using the CTCAE version 5.0 with exception of CRS which will be graded according to adopted grading system in Lee et al, 2014 and TLS that will be graded according to Cairo-Bishop criteria (refer to protocol Appendix 12). Adverse events will be coded using MedDRA.

#### Safety Follow-up

SFU visit will be conducted 30 (+3) days after last administration of AMG 420.

#### **Long-term Follow-up**

LTFU period begin after the SFU visit is completed. The total duration of the LTFU will be up to 5 years from the first dose of AMG 420, or until subject death, whichever is first."

#### 6. Analysis Sets

## 6.1 Safety Analysis Set

Safety Analysis Set defined as all subjects that are enrolled and receive at least 1 dose of AMG 420.

#### 6.2 Dose Limiting Toxicity Evaluable Analysis Set

The analysis of DLT will be restricted to DLT-evaluable subjects. **DLT evaluable**analysis set includes subjects who complete the DLT evaluable period or

experienced a DLT anytime during the DLT evaluable period. A subject will be not

DLT evaluable if he/she drops out before completion of the DLT-evaluable period for

reasons other than a DLT prior to completing the 4 weeks of AMG420 treatment.

The DLT window may also be extended to assess events starting within the window in case the DLT definition is time dependent.

#### 6.3 Pharmacokinetic/Pharmacodynamic Analyses Set(s)

The PK Analysis Set will contain all subjects who have received at least 1 dose of the investigational product and have at least 1 PK sample collected. These subjects will be evaluated for PK analysis unless the number of data points required for analysis is not enough, or significant protocol deviations have affected the data, or if key dosing or sampling information is missing.



Protocol Number: 20160370

**Date:** 12 June 2020 

#### 6.4 Retreatment Analysis Set

Retreatment analysis set defined as subjects that are enrolled and receive at least one dose of AMG 420 during the second course of treatment after attaining CR and subsequently have disease progression while off-therapy.

#### 7. Planned Analyses

#### 7.1 Interim Analysis and Early Stopping Guidelines

#### 7.1.1 Interim Analyses

No specific interim analysis planned.

#### 7.1.2 Dose Level Review Team

DLRT will be responsible for monitoring safety and making recommendations regarding termination of enrollment and dose level/schedule escalation/changes. See Protocol Section 12.3 for further details of DLRT responsibilities.

#### 7.2 Primary Analysis

The primary analysis will occur when the target enrollment is complete and each subject has had the chance to be treated for at least 6 months.

#### 7.3 Final Analysis

A final analysis is planned after all subjects have ended the study.

#### 8. Data Screening and Acceptance

#### 8.1 General Principles

The objective of the data screening is to assess the quantity, quality and statistical characteristics of the data relative to the requirements of the planned analyses. The database will be subject to edit checks outlined in the data management plan (DMP) by Amgen Clinical Data Management (CDM) department. Data inconsistencies and suspicious values will be reviewed and resolved before the database is locked.

#### 8.2 Data Handling and Electronic Transfer of Data

The Amgen Global Study Operations-Data Management (GSO-DM) department will provide all data to be used in the planned analyses. This study will use the RAVE database.

#### 8.3 Handling of Missing and Incomplete Data

The following imputation for missing or incomplete data will be performed if required:

Incomplete adverse event and concomitant medication dates missing data will be imputed as described in Appendix A.



Protocol Number: 20160370

**Date:** 12 June 2020 

Non-pharmacokinetic measurements (eg, biomarker data) that are below the lower limit of quantification will be considered equal to half of the lower limit of quantification for all analyses unless specified otherwise.

#### 8.4 Detection of Bias

Lack of protocol compliance and the potential for biased statistical analyses will be examined by assessing the incidence of important protocol deviations in each cohort. The clinical study team will identify and document the criteria for important protocol deviations.

#### 8.5 Outliers

Outlier data will not be excluded unless scientifically justified.

Pharmacokinetic (PK) serum concentration data will be evaluated for outliers by visual inspection, and decisions to re-assay individual samples will be made in accordance with standard pharmacokinetic evaluation practice.

#### 8.6 Distributional Characteristics

Where appropriate, the assumptions underlying the proposed statistical methodologies will be assessed. If required data transformations or alternative non-parametric methods of analyses will be utilized.

#### 8.7 Validation of Statistical Analyses

Programs will be developed and maintained, and output will be verified in accordance with current risk-based quality control procedures.

Tables, figures, and listings will be produced with validated standard macro programs where standard macros can produce the specified outputs.

The production environment for statistical analyses consists of Amgen-supported versions of statistical analysis software; for example, the SAS System version 9.4 or later.

#### 9. Statistical Methods of Analysis

#### 9.1 General Considerations

Descriptive statistics will be provided for selected demographics, safety, PK, pharmacodynamic and biomarker data by dose, dose schedule, and time as appropriate. Descriptive statistics on continuous data will include means, medians, standard deviations and ranges, while categorical data will be summarized using frequency counts and percentages. Time to event endpoints will be summarized with Kaplan-Meier (KM) proportions at select time points, KM quartiles (when estimable), the number of



Protocol Number: 20160370

**Date:** 12 June 2020 

subjects with events, the number of subjects censored, and censoring reasons. Duration of follow-up for time to event endpoints will be estimated using the reverse Kaplan Meier method (Schemper and Smith, 1996). Point estimates for efficacy endpoints will be accompanied by 2-sided 95% confidence intervals including KM quartiles (Klein and Moeschberger, 1997), KM proportions (Kalbfleisch and Prentice, 1980), and binomial proportions (Clopper and Pearson, 1934). Graphical summaries of the data may also be presented.

#### 9.2 Subject Accountability

The following subject disposition information will be summarized as follows

- Number of screened subjects
- Number of subjects in Safety Analysis Set
- Number (%) of subjects who discontinued treatment
- Number (%) of subjects who discontinued the study
- Primary reason for ending treatment
- Primary reason for study discontinuation

The percentages are based on the number of subjects **enrolled in the study**.

#### 9.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined by the study team before the first subject's initial visit and updated during the IPD reviews throughout the study prior to database lock. These definitions of IPD categories, subcategory codes, and descriptions will be used during the course of the study. Eligibility deviations are defined in the protocol.

#### 9.4 Demographic and Baseline Characteristics

The following descriptive summaries of the demographic and baseline characteristics will be produced: Demographic (ie, age, age groups [< 65, 65-74 and >= 75], sex, race, ethnicity), prior line of therapies (median, range) and baseline characteristics (height, weight, Eastern Cooperative Oncology Group (ECOG) Performance Status will be summarized using descriptive statistics. If multiple races have been reported for a subject, the subject will be categorized as multiple.



Protocol Number: 20160370

**Date:** 12 June 2020 

#### 9.5 Efficacy Analyses

#### 9.5.1 Analyses of Key Secondary Efficacy Endpoint(s)

#### 9.5.1.1 Overall Response Rate

The number (%) of subjects with a best overall response of sCR, CR, VGPR, PR, MR, SD, PD or IE will be summarized.

Overall response rate is defined as the proportion of subjects for whom the best overall response is sCR, CR, VGPR, or PR as determined by International Myeloma Working Group Uniform Response Criteria (IMWG-URC). The ORR along with the associated 95% exact binomial confidence interval (Clopper-Pearson method) will be determined.

#### 9.5.1.2 **Duration of Response**

Kaplan-Meier methods will be used to estimate the distribution of DOR. And the median and other quartiles in addition to the corresponding two-sided 95% confidence intervals will be calculated.

A Kaplan-Meier figure showing the estimated DOR distribution will be provided.

#### 9.5.1.3 MRD Negativity at CR

MRD negativity analysis will be performed for all subjects included in the safety analysis set. Number of MRD[-] responders at CR along with exact 2-sided 95% will be provided by using Clopper & Pearson method

#### 9.5.2 Analyses of Secondary Efficacy Endpoint(s)

#### 9.5.2.1 Progression-free Survival

PFS analysis will be performed for all subjects included in the safety analysis set. The Kaplan-Meier curve will be generated. PFS rate at 3-month intervals and the median and other quartiles in addition to the corresponding two-sided 95% confidence intervals will be provided. Disease progression determined by using IMWG-URC will be used for the analysis.

#### 9.5.2.2 Overall Survival

OS analysis will be performed for all subjects included in the safety analysis set. **The Kaplan-Meier curve will be generated**. Overall survival rate at 3-month intervals, the median and other quartiles in addition to the corresponding two-sided 95% confidence intervals will be calculated.



Protocol Number: 20160370

**Date**: 12 June 2020 

#### 9.5.2.3 Time to Response

Time to response will be calculated for subjects who achieved best overall response of PR, VGPR, CR or sCR. Time to response is calculated as the number of months from the first administration of AMG 420 to the first objective assessment of response (ie, date of the first detection of response) as per IMWG-URC.

Time to response will be descriptively analyzed, summary statistics of the number, mean, standard deviation, median, and range will be reported.

Listings will be produced for all subjects indicating the MRD negativity, OS, PFS, time to response, and duration of response.

#### 9.5.3 Analyses of Exploratory Efficacy Endpoint(s)



## 9.6 Safety Analyses

#### 9.6.1 Analyses of Safety Endpoint(s)

Statistical analyses on safety endpoints will be done using subjects from the Safety Analysis Set (except the analysis of the DLT endpoint, which will be based on subjects from the DLT evaluable set), which includes subjects that are enrolled and received at least 1 dose of AMG 420.

#### 9.6.2 Adverse Events

The Medical Dictionary for Regulatory Activities (MedDRA) version 23.0 or later will be used to code all adverse events to a system organ class and a preferred term. The severity of each adverse event will be graded using CTCAE version 5.0 criteria with exception of CRS which will be graded according to adopted grading system in Lee et al, 2014 and TLS graded according to Cairo-Bishop criteria (refer to protocol Appendix 12). Where appropriate the tables will also be presented by worst grade.

Treatment-emergent adverse events will be summarized based on the number (%) of subjects experiencing events by MedDRA SOC and PT. The denominator for the percentage will be based on the number of subjects in the safety analysis set.



Protocol Number: 20160370

**Date**: 12 June 2020 

#### The subject incidence of adverse events will be summarized for

#### • TEAE

- All treatment-emergent AEs
- Grade 3 or higher treatment-emergent AEs
- Treatment-emergent SAEs
- Treatment-emergent AEs leading to interruption of investigational product
- Treatment-emergent AEs leading to withdrawal of investigational product
- Fatal treatment-emergent AEs

#### Treatment-related AEs

- All treatment-related AEs
- Grade 3 or higher treatment-related AEs
- Treatment-related SAEs
- Treatment-related AEs leading to interruption of investigational product
- Treatment-related AEs leading to withdrawal of investigational product
- Fatal treatment-related AEs

The summaries that are displayed by SOC, PT and grade will be ordered by descending order of incidence of SOC, PT and grade with in each SOC for the total group.

Then summary of TEAEs, summary of TEAEs, TESAEs, Treatment-related TEAEs, and Treatment-related SAEs by SOC, PT and Grade will be generated for extramedullary subjects.

The above adverse event tables will not be created if two or fewer subjects experience the adverse event.

### **Dose Limiting Toxicities**

The analysis of the probability of DLTs will include data from DLT-evaluable subjects (see Protocol Section 7.4.1 for definition of DLT-evaluable). The primary analysis will only include DLTs that occur during the DLT evaluation period. If DLTs occur outside the DLT evaluation period, a sensitivity analysis will be performed where DLTs occurring outside of the specified time interval are included. The number and percentage of subjects reporting DLTs will be evaluated overall and by AMG 420 dose level.



Protocol Number: 20160370

**Date:** 12 June 2020 

## 9.6.3 Laboratory Test Results

Chemistry, Hematology and Coagulation

Actual values and change from baseline for selected chemistry and hematology parameters will be summarized descriptively for each scheduled visit based on the safety analysis set.

| Chemistry | Hematology | Coagulation |
|----------------------|------------|-------------|
| Total bilirubin | ANC | PT or INR |
| ALT (SGPT) | Hemoglobin | APTT |
| AST (SGOT) | Platelets | |
| Alkaline phosphatase | WBC | |
| Creatinine | Lymphocyte | |
| Phosphate | | |
| Calcium (Corrected) | | |
| Potassium | | |
| Sodium | | |
| Albumin | | |
| Glucose | | |
| Amylase | | |
| Lipase | | |

Shift tables will be presented for the baseline toxicity grade by the worst on-study toxicity grade in a table form for selected parameters mentioned above if applicable. CTCAE version 5.0 will be used for toxicity grading for the above mentioned parameters excluding Total bilirubin, ALT (SGPT), AST (SGOT) and Alkaline phosphatase (CTCAE version 4.03 will be used for toxicity grading).

Potential Hy's law cases may be summarized.

#### 9.6.4 Vital Signs

The analyses of vital signs include summary statistics over time and/or changes from baseline over time.

#### 9.6.5 Physical Measurements

The analyses of physical measurements will include summary statistics at baseline.



Protocol Number: 20160370

**Date:** 12 June 2020 

#### 9.6.6 Electrocardiogram

Summaries over time and/or changes from baseline over time will be provided for all ECG parameters. Subjects' maximum post baseline values will be categorized and the number and percentage of subjects in each group will be summarized.



#### 9.6.8 Exposure to Investigational Product

The average dose administration ( $\mu$ g), cumulative dose ( $\mu$ g), number of cycles, duration of treatment, number and percentage of subjects with dose modifications, reasons for modification will be summarized using descriptive statistics. Subject-level data may be provided instead of the summary if the subject incidence is low or single dose is given.

Descriptive statistics will be produced to describe the exposure to investigational product by treatment group.

Extent of exposure to study treatments will be summarized for Safety population

- Duration of treatment (days)
  - Defined as the duration (in weeks) from the date of the first dose to the date of the last dose of study drug + 1
- Total number of treatment cycles started
  - Defined as the total number of treatment cycles in which at least one dose of study drug is administered.
- Cumulative dose received of AMG420 across all cycles, defined as the cumulative dose of AMG 420.
- Average dose of AMG420, defined as the total dose received divided by the number of days on treatment administered.

#### 9.6.9 Exposure to Concomitant Medication

Number and proportion of subjects receiving therapies of interest will be summarized by preferred term for each treatment group as coded by the World Health Organization Drug dictionary.

#### 9.7 Other Analyses

#### 9.7.1 PK Analyses

The PK parameters of AMG 420 including, but not limited to, average  $C_{ss}$ , clearance, and half-life ( $t_{1/2}$ ) for serum AMG 420 will be estimated using non-compartmental methods and summarized by dose level using means, geometric means, standard



Protocol Number: 20160370

**Date**: 12 June 2020 

deviations, coefficients of variation, medians, minimums, and maximums. Individual concentration-time profiles will be summarized by dose level. Plasma AMG 420 concentrations at each time point along with PK parameter values may be listed for each subject. Summary statistics will be computed for each sampling time and parameter as appropriate. The relationship between AMG 420 exposure and efficacy/safety may be conducted.

## 9.7.2 Analyses of Pharmacokinetic or Pharmacokinetic/Pharmacodynamic Endpoints

PK/PD analyses will be provided by the Department of Clinical Pharmacology, Modeling & Simulation (CPMS). Actual collection times of PK samples will be recorded to assess the plasma concentration. The PK parameter estimates for AMG420 will be summarized. Exploratory analyses may be performed to evaluate the relationship between the estimated PK parameters and selected safety, biomarker, or clinical effect endpoints. In addition, the population modeling program may be used to fit a nonlinear mixed effects model to estimate PK parameters. Details regarding the analyses will be provided in a separate analysis plan by CPMS.

#### 9.7.3 Analyses of Clinical Outcome Assessments

Analysis of clinical outcome assessments is not planned for this study.

### 9.7.4 Analyses of Health Economic Endpoints

Analyses of Health Economic Endpoints are not planned for this study.

## 9.7.5 Analyses of Biomarker Endpoints

The analysis of Biomarker will be described and performed by Clinical Biomarker Group.

#### 10. Changes From Protocol-specified Analyses

There are no changes to the protocol-specified analyses.



Protocol Number: 20160370

**Date:** 12 June 2020 

#### 11. Literature Citations / References

Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of the binomial. *Biometrika*. 1934;26(4):404-413.

Ji Y, Liu P, Li Y, Bekele BN. A modified toxicity probability interval method for dose-finding trials. *Clin Trials*. 2010;7(6):653-663.

Kalbfleisch JD, Prentice RL. The Statistical Analysis of Failure Time Data, Hoboken, New Jersey: John Wiley & Sons; 1980.

Klein JP, Moeschberger ML. Survival Analysis: Techniques for Censored and Truncated Data, New York: Springer-Verlag; 1997.

Kumar S, Paiva B, Anderson KC, et al. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. *Lancet Oncol.* 2016;17(8):e328-346.

Schemper M, Smith TL. A note on quantifying follow-up in studies of failure time. *Control Clin Trials.* 1996;17(4):343–46.

Lee JJ, Liu DD. A predictive probability design for phase II cancer clinical trials. *Clinical Trials*. 2008;5(2):93-106.

Thall P, Simon R, Estey E. Bayesian sequential monitoring designs for single-arm clinical trials with multiple outcomes *Statistics in Medicine*. 1995;14:357-379



**Protocol Number:** 20160370

**Date:** 12 June 2020 

## 12. Prioritization of Analyses

No Priority of outputs planned for this study

## 13. Data Not Covered by This Plan

The analysis of Biomarkers (except MRD) is not covered in this plan.



**Protocol Number:** 20160370

**Date:** 12 June 2020 

## 14. Appendices



Protocol Number: 20160370

**Date:** 12 June 2020 

#### Appendix A. Reference Values/Toxicity Grades

The Common Terminology Criteria for Adverse Events (CTCAE) v5.0 is available at the following link:

http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm

# <u>Technical Detail and Supplemental Information Regarding Statistical Procedures</u> <u>and Programs</u>

Imputation Rules for Partial or Missing Stop Dates

If the month and year are present, impute the last day of the month. If only the year is present, impute December 31 of that year. If the stop date is entirely missing, assume the event or medication is ongoing.

Imputation Rules for Partial or Missing Start Dates

| | Stop Date | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | Com <sub>l</sub> | olete:<br>nmdd | Partial: | yyyymm | Partial: yyyy | | |
| Start<br>Date | | <1st | ≥1 <sup>st</sup> | <1st | ≥1 <sup>st</sup> Dose | <1st | ≥1 <sup>st</sup> Dose | Minaina |
| Date | 4 ct | Dose | Dose | yyyymm | yyyymm | уууу | уууу | Missing |
| Partial: | =1 <sup>st</sup><br>Dose<br>yyyymm | N/A | 1 | N/A | 1 | N/A | 1 | 1 |
| yyyymm | ≠ 1 <sup>st</sup> Dose yyyymm | | 2 | 2 | 2 | 2 | 2 | 2 |
| Partial: | =1 <sup>st</sup> Dose yyyy | N/A | 1 | N/A | 1 | N/A | 1 | 1 |
| уууу | ≠ 1 <sup>st</sup> Dose уууу | | 3 | | 3 | 3 | 3 | 3 |
| Mis | sing | 4 | 1 | 4 | 1 | 4 | 1 | 1 |

<sup>1 =</sup> Impute the date of first dose



<sup>2 =</sup> Impute the first day of the month

<sup>3 =</sup> Impute January 1 of the year

<sup>4 =</sup> Impute January 1 of the stop year

Protocol Number: 20160370

**Date**: 12 June 2020 

Note: For subjects who were never treated (first dose date is missing), partial start dates will be set to the first day of the partial month.

Note: If the start date imputation leads to a start date that is after the stop date, then do not impute the start date.

Imputation rules for stop date:

For partial stop date mmyyyy, impute the last day of the month.

For partial stop date yyyy, impute December 31 of the year.

For completely missing stop date, do not impute.

If the stop date imputation leads to a stop date that is after the death date, then impute the stop date as the death date.

If the stop date imputation leads to a stop date that is before the start date, then there is a data error and do not impute the stop date. (ie. set the stop date as missing).

#### **Code Fragments:**

Provisional Code Fragments for calculating a confidence interval using the Clopper Pearson Method. The following example SAS code will be utilized for the response rate analysis providing the proportion of subjects responding to treatment with corresponding 80% confidence intervals.

```
data propci (keep = ns p low_ci upp_ci);
n=xx; * total n within the treatment group;
do ns= xx; *number of responders;
p=ns/n; * response rate;
q=1-p;
lowF=FINV(0.1, 2*ns, 2*(n-ns+1)); /* use for 2-sided 80% CI */
UppF=FINV(1-0.1, 2*(ns+1), 2*(n-ns)); /* use for 2-sided 80% CI */
low_ci = 1 / (1+(n-ns+1) / (ns*lowf)); * lower CI for response rate;
upp_ci = 1 / (1+(n-ns) / ((ns+1)*uppf)); *upper CI for response rate;
if p=1 then upp_ci=1;
if p=0 then low_ci =0;
output;
end;run;
```



**Protocol Number:** 20160370

**Date:** 12 June 2020 

## Appendix B. Guidance for Response Confirmation

For responses assessed by investigator, the following table and notes will be used to confirm the responses:

# Confirmation of Response Assessed by Investigator at Each Visit (applicable to MR or better and PD)

| "Has response been confirmed" Entered on IMWG Response CRF for the current assessment (Yes/No) | 'Has response<br>been confirmed'<br>Entered on<br>IMWG Response<br>CRF for the next<br>assessment<br>(Yes/No) | Response Category of the current and the next assessments | Confirmation of the current assessment |
|---|---|---|---|
| Yes | - | - | Confirmed |
| No | Yes | If the current assessment is MR or better, and the next assessment is no worse than the current one, keep the current response status as is. | Confirmed |
| | | If the current assessment is MR or better, and the next assessment is worse than the current one but also is MR or better, select the response status same as the next assessment. | Confirmed |
| | | If the current assessment is PD, and the next assessment is also PD, keep the current response status as is. | Confirmed |
| | | If the current assessment is PD, but the next assessment is not PD, keep the current response status as is. | Unconfirmed |
| | No | Leave the response as is. | Unconfirmed |



**Protocol Number: 20160370** 

**Date:** 12 June 2020 

#### Note:

Response assessments done after initiation of new anti-cancer therapy will be excluded. But if new anti-cancer therapy is started before confirmed progressive disease, additional testing during subsequent therapy can be used to confirm progressive disease (PD), as long as this testing is within 35 days from the last disease assessment on study.

Stable disease (SD) means the response does not fulfil criteria for a confirmed MR, PR, VGPR, CR, sCR, or PD. An assessment of SD does not need to be confirmed, however it should be remains same at least 6 weeks. A response of SD is not upgraded until there is a confirmed response of sCR, CR, VGPR, PR, MR or PD.

For subjects that do not qualify for a confirmed response or stable disease (SD), the BOR will be not evaluable



**Protocol Number:** 20160370

**Date:** 12 June 2020 

## Appendix C. Clinical Outcome Assessment Forms/Instruments

Not applicable



**Protocol Number:** 20160370

**Date:** 12 June 2020 

## Appendix D. Health Economic Forms/Instruments

Not applicable



**Protocol Number:** 20160370

**Date:** 12 June 2020 

## Appendix E. Details of PK or PK/PD Methods for Modeling

CPMS group will be responsible for PK/PD modeling.

